CLINICAL TRIAL: NCT01296100
Title: DEMOnstration Area for Primary Prevention of Type 2 Diabetes, JUAN Mina and Barranquilla, Colombia
Brief Title: DEMOJUAN- DEMOnstration Area for Primary Prevention of Type 2 Diabetes, JUAN Mina and Barranquilla, Colombia
Acronym: DEMOJUAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigacion Sanitaria (Network)
Collaborators: International Diabetes Federation (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LT09-258
Record Dates: First submitted 2011-02-12; First posted 2011-02-15 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes; Glucose Metabolism Disorders
Keywords: impaired glucose tolerance; nutrition; physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Glucose Intolerance; Motor Activity | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (nutrition) (Experimental): The 200 study participants of this arm will first receive 6 months of nutritional counseling and thereafter combined nutrition/physical activity counseling during 18 month. The counseling sessions consists of monthly group seminars (10 participants/group) and totally 6 individual visits with a nutritionist and 6 visits with a physical activity expert.
  Interventions: Behavioral: Lifestyle intervention (nutrition)
- Lifestyle counseling (physical activity) (Experimental): The 200 study participants of this arm will first receive 6 months of physical activity counseling and thereafter combined nutrition/physical activity counseling during 18 month. The counseling sessions consists of monthly group seminars (10 participants/group) and totally 6 individual visits with a nutritionist and 6 visits with a physical activity expert.
  Interventions: Behavioral: Lifestyle intervention (physical activity)

INTERVENTIONS:
Behavioral: Lifestyle intervention (nutrition) — The 200 study participants of this arm will first receive 6 months of Nutritional counseling and thereafter combined nutrition/physical activity counseling during 18 month. The counseling sessions consists of monthly group seminars (10 participants/group) and totally 6 individual visits with a nutritionist and 6 visits with a physical activity expert.
  Arms: Lifestyle intervention (nutrition)
Behavioral: Lifestyle intervention (physical activity) — The 200 study participants of this arm will first receive 6 months of physical activity counseling and thereafter combined nutrition/physical activity counseling during 18 month. The counseling sessions consists of monthly group seminars (10 participants/group) and totally 6 individual visits with a nutritionist and 6 visits with a physical activity expert.
  Arms: Lifestyle counseling (physical activity)

SUMMARY:
The main aim of this study is to investigate to what extent it is possible to reach normal glucose metabolism and optimal cardiovascular disease (CVD) risk factor levels with early lifestyle interventions in people at high risk of type 2 diabetes compared with those who receive standard therapy (usual care) only.

The project will show the effect of these interventions for the first time in people of low socio-economic levels living in a Caribbean environment.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is one of the fastest growing public health problems in both developed and developing countries. The development of T2D is a slow process and involves both genetic and environmental effects. It is commonly agreed that T2D may develop only in people that carry a genetic predisposition to the disease. Based on epidemiological observations about half of the people will develop T2D during their lifetime, and up to 30-35% will have IGT. Therefore, it is likely that more than half of the population carry genes that predispose the development of T2D. In people genetically predisposed to the disease, the probability to develop T2D is very high once exposed to unhealthy lifestyles such as obesity, unbalanced diet and physical inactivity. While we cannot change the genes, the only way to prevent T2D and its serious complications is the modification of lifestyle risk factors. Therefore, it is very important to understand the role of preventive lifestyle intervention as a key treatment in T2D prevention. Once established, T2D is difficult to treat. Despite pharmacologic treatment blood glucose levels trend to increase over time. Thus, the most efficient way to manage T2D is to prevent diabetes from developing. Also complications of T2D can best be postponed by postponing the onset of the primary disease itself. The efforts to prevent the disease need to start as early as possible and address all susceptibility factors. Fortunately, recent studies have convincingly demonstrated that prevention of T2D is possible. This project will show for the first time how lifestyle interventions work in people with IGT in the Caribbean population. The results of this study will be sued for policy making and planning of primary prevention activities not only in the local health-care system but in the entire Caribbean region.

ELIGIBILITY:
Inclusion Criteria:

* 34-69 years-of-age with diagnosed IGT
* Informed consent given.

Exclusion Criteria:

* Patients with pharmacologically-treated diabetes
* Hypertriglyceridaemia under drug treatment
* History of life-limiting diseases or events
* Unwillingness to sign the informed consent.

Ages: 34 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who reach normal levels of all glycaemic parameters. | Month 24 of the intervention
  * Proportion of patients whose fasting glucose level is less than 6.1 mmol/l
  * Proportion of patients whose 2-hour glucose level is less than 7.8 mmol/l

SECONDARY OUTCOMES:
Difference in reduction of 10 year-estimated cardiovascular risk score of 10% between the standard therapy control group and the lifestyle intervention groups (WHO CVD prediction chart). | Month 24 of the intervention
  * Proportion of patients whose blood pressure level is less than 130/80 mmHg
  * Proportion of patients whose serum HDL cholesterol level is more than 1.2 mmol/l
  * Proportion of patients whose serum LDL cholesterol level is less than 2.0 mmol/l
  * Proportion of patients whose total/HDL cholesterol ratio is less than 4.0
  * Proportion of patients whose weight reduction is more than 5%

CONTACTS AND LOCATIONS:
Overall Officials: Jaakko O Tuomilehto, MD, PhD, Principal Investigator — University of Helsinki; Tania Acosta, MD, Study Chair — CIIS LTDA; Noël C Barengo, MD, PhD, MPH, Study Chair — CIIS LTDA; Astrid Arrieta, MD, Study Director — CIIS LTDA; Carlos Ricaurte, Study Chair — CIIS LTDA
Locations (5):
- Colombia (5):
  - Camino Bosques de María, Barranquilla, Barranquilla
  - Camino Sur Occidente El Pueblo, Barranquilla, Barranquilla
  - Centro de INvestigacion Sanitaria, Barranquilla, Barranquilla
  - Paso Las Malvinas, Barranquilla, Barranquilla
  - Paso Nueva Era, Barranquilla, Barranquilla

IPD SHARING:
Plan to Share IPD: Yes
The study group is ready to share the data in de-identified format once the main results have been reported or in case any journal may ask for the data to run a check.

REFERENCES:
- [Background] Schwarz PE, Li J, Lindstrom J, Tuomilehto J. Tools for predicting the risk of type 2 diabetes in daily practice. Horm Metab Res. 2009 Feb;41(2):86-97. doi: 10.1055/s-0028-1087203. Epub 2008 Nov 19. PMID 19021089
- [Background] Lindstrom J, Peltonen M, Eriksson JG, Aunola S, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS) Group. Determinants for the effectiveness of lifestyle intervention in the Finnish Diabetes Prevention Study. Diabetes Care. 2008 May;31(5):857-62. doi: 10.2337/dc07-2162. Epub 2008 Feb 5. PMID 18252900
- [Background] Lindstrom J, Louheranta A, Mannelin M, Rastas M, Salminen V, Eriksson J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. The Finnish Diabetes Prevention Study (DPS): Lifestyle intervention and 3-year results on diet and physical activity. Diabetes Care. 2003 Dec;26(12):3230-6. doi: 10.2337/diacare.26.12.3230. PMID 14633807
- [Derived] Acosta T, Barengo NC, Arrieta A, Ricaurte C, Tuomilehto JO. A demonstration area for type 2 diabetes prevention in Barranquilla and Juan Mina (Colombia): Baseline characteristics of the study participants. Medicine (Baltimore). 2018 Jan;97(1):e9285. doi: 10.1097/MD.0000000000009285. PMID 29505512
- See also: Related Info — http://www.idfbridges.org/projects/1/4